CLINICAL TRIAL: NCT01427296
Title: A Phase 4, Randomized, Active Comparator, Open-Label, Multicenter Study to Assess the Safety and Efficacy of OsmoPrep® Tablets Versus HalfLytely® and Bisacodyl Tablet Bowel Prep Kit for Colon Cleansing
Brief Title: Safety and Efficacy of OsmoPrep® Tablets Versus HalfLytely® and Bisacodyl Tablet Bowel Prep Kit for Colon Cleansing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSBP4011
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Colon Cleansing
Keywords: Colon Cleansing; Bowel Prep; Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OsmoPrep Tablets (Active Comparator)
  Interventions: Drug: Oral sodium phosphate solution
- HalfLytely and Bisacodyl Tablet (Active Comparator)
  Interventions: Drug: Polyethylene glycol

INTERVENTIONS:
Drug: Polyethylene glycol — HalfLytely and Bisacodyl Tablet Bowel Prep Kit, administered as 1 bisacodyl tablet followed by HalfLytely oral solution in a total liquid volume of approximately 2 L
  Arms: HalfLytely and Bisacodyl Tablet
Drug: Oral sodium phosphate solution — OsmoPrep tablets (48 g), administered as 32 total tablets in a total liquid volume of approximately 2 L
  Arms: OsmoPrep Tablets

SUMMARY:
The purpose of this study is to compare the safety and efficacy of OsmoPrep tablets versus HalfLytely and Bisacodyl Tablet Bowel Prep Kit in subjects who are undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age, inclusive
* Scheduled for colonoscopy within 21 days of the screening visit
* Able to swallow tablets the size of a multivitamin without difficulty

Exclusion Criteria:

* History of biopsy-proven acute phosphate nephropathy
* Known allergy or hypersensitivity to treatment arms
* History of gastric stapling or bypass procedure or history of gastric retention
* History of any other sodium phosphate preparation within 6 months prior to colonoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2154 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2014-03-11 (Actual); Study Completion 2014-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - San Carlos, California
  - Bristol, Connecticut
  - Macon, Georgia
  - Suwanee, Georgia
  - Hagerstown, Maryland
  - Wyoming, Michigan
  - Mexico, Missouri
  - Vineland, New Jersey
  - Great Neck, New York
  - New York, New York
  - Fayetteville, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Mentor, Ohio
  - Plano, Texas
  - Chesapeake, Virginia
  - Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OsmoPrep Tablets | HalfLytely and Bisacodyl Tablet
Started | 1041 | 1051
Completed | 1041 | 1051
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OsmoPrep Tablets | HalfLytely and Bisacodyl Tablet | Total
Number analyzed (Participants) | 1041 | 1051 | 2092
Age, Customized [Count of Participants; unit: Participants]
  <65 | 906 | 932 | 1838
  >=65 | 135 | 119 | 254
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 616 | 645 | 1261
  Male | 425 | 406 | 831

OUTCOME MEASURES:

1. Primary Outcome: Distribution of the Overall Colon-cleansing Scale in Each Treatment Group.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | OsmoPrep Tablets | HalfLytely and Bisacodyl Tablet
Number analyzed (Participants) | 1032 | 1040
Participants
  Excellent | 618 | 243
  Good | 275 | 423
  Fair | 116 | 286
  Inadequate | 23 | 88

ADVERSE EVENTS:
Arm/Group | OsmoPrep Tablets | HalfLytely and Bisacodyl Tablet
Serious Adverse Events (participants affected / at risk) | 20/1041 | 19/1051
Other Adverse Events (participants affected / at risk) | 443/1041 | 352/1051
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OsmoPrep Tablets (N=1041) | HalfLytely and Bisacodyl Tablet (N=1051)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic Fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Bladder perforation (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OsmoPrep Tablets (N=1041) | HalfLytely and Bisacodyl Tablet (N=1051)
Abdominal pain (Gastrointestinal disorders) | 12 | 21
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhea (Gastrointestinal disorders) | 10 | 12
Gastritis (Gastrointestinal disorders) | 21 | 11
Nausea (Gastrointestinal disorders) | 42 | 50
Oesophagitis (Gastrointestinal disorders) | 10 | 7
Vomiting (Gastrointestinal disorders) | 23 | 45
Brochitis (Infections and infestations) | 18 | 15
Nasopharyngitis (Infections and infestations) | 9 | 20
Sinusitis (Infections and infestations) | 18 | 19
Upper respiratory tract infection (Infections and infestations) | 24 | 25
Urinary tract infection (Infections and infestations) | 34 | 38
Hyperphosphataemia (Metabolism and nutrition disorders) | 136 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 21
Headache (Nervous system disorders) | 20 | 16
Haematuria (Renal and urinary disorders) | 8 | 15
Proteinuria (Renal and urinary disorders) | 14 | 9
Hypertension (Vascular disorders) | 15 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes